CLINICAL TRIAL: NCT03333330
Title: Non Invasive Vascular Imaging Combined With Systemic Biomarkers and Brain Magnetic Resonance Imaging for Identification of Asymptomatic Patients With Unstable Carotid Atherosclerosis
Brief Title: IMaging Della PLAcca Carotidea
Acronym: IMPLAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Enrico Ammirati (Other)
Responsible Party: Sponsor-Investigator, Enrico Ammirati, Principal Investigator of the grant number GR-2009-1608780 funded by the Italian Ministry of Health Grant, Università Vita-Salute San Raffaele
Organization: Università Vita-Salute San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GR-2009-1608780
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Carotid Artery Plaque; Atherosclerosis; Ischemic Stroke
Keywords: Carotid atherosclerosis; Carotid plaque; Brain magnetic resonance imaging; Contrast enhanced ultrasound; Carotid CT angiography; Silent brain ischemia; Vascular cognitive impairment
MeSH Terms: conditions — Carotid Stenosis; Atherosclerosis; Ischemic Stroke; Carotid Artery Diseases | interventions — contrast agent BR1; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid imaging with Visipaque 320 and SonoVue (Experimental): Patients undergo to brain MRI, carotid contrast-enhanced CTA, duplex ultrasound, CEUS, blood sampling, clinical structured interview.
  Intervention is related to the administration of contrast agents:
  Visipaque 320 for contrast-enhanced CTA, and SonoVue for CEUS
  Interventions: Drug: Visipaque 320 and SonoVue

INTERVENTIONS:
Drug: Visipaque 320 and SonoVue — Intervention is related to the administration of contrast agents:
  Iodixanol, 320 mg of iodine per millilitre, Visipaque 320 (GE Healthcare, Milwaukee, WI, USA) for contrast-enahnced CTA, Sodium hexafluoride (SonoVue, Bracco Imaging, Milan, Italy) for CEUS
  Other Names: Contrast agents

SUMMARY:
Background-White matter hyperintensities (WMH), patchy areas of hyperintense signal on T2-weighted or Fluid Attenuated Inversion Recovery sequences on brain magnetic resonance imaging (MRI), are believed to reflect cerebral burden of ischemic damage and are associated to incident stroke, dementia and eventually mortality in otherwise healthy subjects. Also brain atrophy has been related with presence of carotid atherosclerosis and vascular cognitive impairment. Carotid atherosclerosis may contribute to the genesis of WMH. A recent meta-analysis by our group comprising 5306 subjects was able to demonstrate an association between the presence of carotid atherosclerosis and WMH (odds ratio, OR, 1.42, 95% confidence interval [CI] 1.22-1.66).

Objective-To evaluate the relation between carotid artery plaque characteristics, cardiovascular risk factors and brain atrophy/WMH burden analyzed quantitatively as number and volume of lesions and as brain volumes, and progression over 18 months of follow up in subjects asymptomatic for cerebrovascular disease with a carotid artery stenosis <70%.

DETAILED DESCRIPTION:
* Ischemic stroke and vascular cognitive impairment pose a massive clinical, social and economic burden. Disruption of carotid plaques, often non-obstructive, with subsequent thrombosis and distal embolization is one of leading pathogenetic mechanism of ischemic stroke. The widespread use of brain magnetic resonance imaging (MRI) has enabled an increased recognition, especially in elderly subjects, of cerebral alterations in apparently healthy individuals.
* Carotid plaque may be causative in the development of white matter hyperintensities (WMH, patchy areas of signal hyperintensity on T2-weighted and/or fluid attenuated inversion recovery -FLAIR- sequences), silent brain infarcts (SBI) and eventually brain atrophy.
* The hypothesis of the investigators is that carotid plaques with features of vulnerability detected by multimodality imaging (including standard ultrasound, contrast enhanced ultrasound -CEUS-, contrast enhanced CT angiography) and larger extent of atherosclerotic process, even if determining only an intermediate degree of stenosis, could bear a more rapid progression of silent WMH and brain atrophy.
* Carotid CT and CEUS allow fast and reproducible evaluation of plaque size and morphology, alongside with functional parameters. Plaque density and positive remodelling on CT have been repeatedly associated to histological features of plaque vulnerability. At the same time, when compared to standard duplex evaluation, CEUS allowed a better imaging definition of plaque margins and extension, and to evaluate intraplaque neovascularization. The latter associates with local inflammation and plaque vulnerability, and might give rise to plaque hematomas, which are among the substrates for lesion progression and for the development of atherothrombosis.
* In the initial phase of the study also hybrid imaging with positron tomography and computed tomography angiography (PET/CTA) using 11C-PK11195 was used to detect and quantify intraplaque inflammation in humans.(7) C-PK11195 is a selective ligand for translocator protein, 18kDa (TSPO), which is highly expressed on the surface of activated monocytes/macrophages. This part of the study was prematurely stopped due to problems with the production of the radiotracer with 11[C] (only 13 patients were studied with this approach).

Primary endpoints:

- The primary endpoint is to identify independent predictors (plaque-related or patient-related) with the progression of WMH through multivariable logistic regression analysis.

Progression of WMH was considered as dichotomous variable: progression versus no progression of WMH.

- The co-primary end-point is to identify independent predictors (plaque-related or patient-related) with the progression of gray matter (GM)/all brain atrophy through multivariable logistic regression analysis. Progression of brain atrophy was considered as dichotomous variable: progression versus no progression of GM/all brain atrophy.

Statistical considerations:

The investigators calculated the sample size for multivariate logistic regression analysis with a power of 0.8 and an alpha of 0.05. The investigators will analyze the highest tertile of carotid plaques burden in terms of plaque volume versus others (see Sillesen, 2012). By definition, the prevalence of high burden atherosclerosis will be 33%. The investigators estimated a clinically relevant probability of progressing in terms of WMH in the high burden group to be 50%, while subjects without high burden plaques are estimated to progress in terms of WMH as the general population with carotid atherosclerosis in a similar time frame. This probability would be estimated to be around 15% (see Dufoil, 2005 and Pico, 2002). The estimated sample size would be 58 individuals.

ELIGIBILITY:
Inclusion Criteria:

- bearing an asymptomatic carotid stenosis of 30-70% in diameter, as established by Doppler-measured peak systolic flow velocity, according to the Society of Radiologists in Ultrasound Consensus Conference (Grant et al. Radiology 2003).

Exclusion Criteria:

* pregnancy or possibility of pregnancy,
* history of allergic diathesis,
* history of stroke or transitory ischemic attack,
* previous carotid artery stenting or carotid endarterectomy,
* history of autoimmune vasculitis,
* History of drug abuse, alcohol abuse or any psychiatric or social condition which may contraindicate the participation to a clinical study
* life expectancy of less than 18 months due to underlying medical conditions,
* presence of cognitive impairment preventing the patient from providing informed consent,
* Atrial fibrillation or previous cardiac surgery or positioning of intracardiac devices (excluded coronary stents) as potential confounding causes of cerebral ischemic damage,
* Known patent foramen ovale (PFO) necessitating anti-platelet treatment
* Current anti-coagulation,
* Previous infections to the central nervous system (CNS)
* Previous surgery to the CNS
* History of anoxic damage to the CNS
* Dementia
* Contraindications to computed tomography angiography (CTA, estimated Glomerular Filtration Rate<60 mL/min; history of allergic reaction to iodinated contrast media),
* Specific contraindication to MRI:

  * Claustrophobia
  * Sickle cell anemia
  * Systemic mastocytosis
  * Implanted cardiac devices (i.e. pacemakers, implantable cardioverter defibrillators)
  * Vascular clips
  * Vertebral distractors
  * Infusion pumps
  * Neurostimulators
  * Liquor derivations
  * Any device which could be dispositioned in the presence of a strong magnetic field

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Changes of total cerebral white matter lesions from baseline (T2-weight lesions, in terms of number and total volumes indexed to the total brain volume) | 18 months
  We expect that asymptomatic patients with carotid atherosclerosis with characteristics of vulnerability of the plaque can develop a larger burden of silent cerebral ischemic lesions along the timeframe of the study. We are going to compare patients with progression compared those without significant progression or no progression.

SECONDARY OUTCOMES:
Changes of total brain volume and grey matter volume from baseline | 18 months
  We expect that asymptomatic patients with carotid atherosclerosis with characteristics of vulnerability of the plaque can develop atrophy of the total brain volume or/and grey matter volume along the timeframe of the study. We are going to compare patients with progression of atrophy compared those without significant progression or no progression.
Changes of ipsilateral cerebral white matter lesions from baseline (T2-weight lesions, in terms of number and total volumes indexed to the total brain volume) | 18 months
  We expect that asymptomatic patients with carotid atherosclerosis with characteristics of vulnerability of the plaque can develop a larger burden of silent cerebral ischemic lesions along the timeframe of the study. We are going to compare patients with progression compared those without significant progression or no progression.
Changes of the carotid total plaque area and extent of CEUS positive plaques | 18 months
  We expect that asymptomatic patients with carotid atherosclerosis with characteristics of vulnerability of the plaque based on CEUS positive plaques and based on cardiovascular risk factors and ongoing treatments can develop a larger extent of total plaque area or/and extent of CEUS positive plaque.
Compare the esteem of the degree and the characteristics of the main plaque with standard Duplex scan versus CEUS using contrast enhanced carotid CT scan as gold standard | at baseline
  We expect that CEUS can be superior compared with standard Duplax scan of the carotid artery in the evaluation of degree of stenosis and presence of irregularity on the surface of the plaque.

OTHER OUTCOMES:
Specific biomarkers (specific T-cell subsets and monocytic subsets and other cytokines) can be associated with WMH and brain atrophy at base line and at follow up (biomarkers to identify progression of WMHs and brain atrophy) | 18 months
  We expect in particular that circulating HLA-DR+CD4+T cells and CD14+CD16- monocytes will be increased in patients with WMH and/or brain atrophy progression

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ammirati, Doctor, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda and Università Vita-Salute San Raffaele; both in Milan, Italy; Paolo G Camici, Professor, Study Chair — Università Vita-Salute San Raffaele and Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ammirati E, Moroni F, Magnoni M, Rocca MA, Messina R, Anzalone N, De Filippis C, Scotti I, Besana F, Spagnolo P, Rimoldi OE, Chiesa R, Falini A, Filippi M, Camici PG. Relation between characteristics of carotid atherosclerotic plaques and brain white matter hyperintensities in asymptomatic patients. Sci Rep. 2017 Sep 5;7(1):10559. doi: 10.1038/s41598-017-11216-x. PMID 28874779
- [Result] Ammirati E, Moroni F, Magnoni M, Di Terlizzi S, Villa C, Sizzano F, Palini A, Garlaschelli K, Tripiciano F, Scotti I, Catapano AL, Manfredi AA, Norata GD, Camici PG. Circulating CD14+ and CD14highCD16- classical monocytes are reduced in patients with signs of plaque neovascularization in the carotid artery. Atherosclerosis. 2016 Dec;255:171-178. doi: 10.1016/j.atherosclerosis.2016.10.004. Epub 2016 Oct 6. PMID 27751505
- [Result] Ammirati E, Magnoni M, Moroni F, Di Terlizzi S, Scotti I, Villa C, Sizzano F, Impellizzeri M, Fanelli G, Esposito G, Chiesa R, Camici PG. Reduction of Circulating HLA-DR+ T Cell Levels Correlates With Increased Carotid Intraplaque Neovascularization and Atherosclerotic Burden. JACC Cardiovasc Imaging. 2016 Oct;9(10):1231-1233. doi: 10.1016/j.jcmg.2015.10.010. Epub 2016 Jan 6. No abstract available. PMID 26777226
- [Result] Moroni F, Magnoni M, Vergani V, Ammirati E, Camici PG. Fractal analysis of plaque border, a novel method for the quantification of atherosclerotic plaque contour irregularity, is associated with pro-atherogenic plasma lipid profile in subjects with non-obstructive carotid stenoses. PLoS One. 2018 Feb 12;13(2):e0192600. doi: 10.1371/journal.pone.0192600. eCollection 2018. PMID 29432486
- [Derived] Ammirati E, Moroni F, Magnoni M, Rocca MA, Anzalone N, Cacciaguerra L, Di Terlizzi S, Villa C, Sizzano F, Palini A, Scotti I, Besana F, Spagnolo P, Rimoldi OE, Chiesa R, Falini A, Filippi M, Camici PG. Progression of brain white matter hyperintensities in asymptomatic patients with carotid atherosclerotic plaques and no indication for revascularization. Atherosclerosis. 2019 Aug;287:171-178. doi: 10.1016/j.atherosclerosis.2019.04.230. Epub 2019 May 6. PMID 31101367

DOCUMENTS (2):
  • Study Protocol (2012-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03333330/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03333330/SAP_001.pdf